CLINICAL TRIAL: NCT00977899
Title: Malaria Transmission-Blocking Pfs25-Pfs25 Conjugate Vaccine
Brief Title: Phase 1 Study of the Safety and Immunogenicity of a Malaria Transmission-blocking Pfs25-Pfs25 Conjugate Vaccine
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 090213; 09-CH-0213
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2013-03-05

CONDITIONS: Malaria; Malaria Vaccines; Plasmodium Falciparum Malaria
Keywords: Plasmodium Falciparum; Alum Adsorbed; Ookinete Surface Protein; Malaria Vaccine; Healthy Volunteer; HV
MeSH Terms: conditions — Malaria; Malaria, Falciparum

INTERVENTIONS:
Biological: Malaria Transmission-Blocking Pfs25-Pfs25 Conjugate Vaccine

SUMMARY:
Background:

* Malaria, a disease transmitted by mosquitoes, affects millions of people with the highest frequency, morbidity, and mortality in infants and young children. Plasmodium falciparum and Plasmodium vivax, the most common and severe forms of malaria, have host- and stage-specific proteins that can induce immunity to the disease.
* Vaccines against stages that infect mosquitoes will prevent the spread of malaria. Researchers have developed a vaccine composed of a single protein, Pfs25, to induce antibodies in the human host that will be ingested by the mosquito and prevent the malaria parasite from reproducing and stop transmission of the disease. Because Pfs25 is present only in the mosquito, humans do not develop antibodies to this antigen even in endemic areas. Repeated injections of this vaccine may be necessary.

Objectives:

- To establish the safety and optimal dosage of a malaria vaccine developed with the Pfs25 protein.

Eligibility:

- Healthy adults between 18 and 49 years of age who have never had malaria or received a malaria vaccine.

Design:

* Two doses of Pfs25 conjugate (10 micrograms and 25 micrograms) will be evaluated in this study. Participants will receive only one of these doses in order to provide the best scientific data for evaluation.
* To determine eligibility, participants will provide a medical history and have a physical examination, and will provide blood and urine samples to test for HIV/AIDS, hepatitis, and other conditions that would prevent them from participating.
* Eligible participants will receive one injection of the vaccine. The injection will be followed 30 minutes later with a temperature reading and an inspection of the vaccine site.
* Upon leaving the clinic, participants will receive diary forms, a digital thermometer, a ruler, and instructions about how to take their temperature and to measure redness and swelling (if any) at the injection site. About 6 hours later, and daily for 3 days, participants will take their temperature at home and examine the injection site. Participants will be examined at the clinic at 48 to 72 hours and on day 7 after an injection. A blood sample will be taken 1 week after immunization. - Participants will receive a second and third injection of the same vaccine at 6-week intervals, and will follow the same recording procedure given above. Further blood samples will be taken at regular intervals for up to 12 months after the vaccination, as directed by the study researchers.

DETAILED DESCRIPTION:
Malaria is a disease affecting millions of people in Africa, Asia, Central and South America . It has its highest frequency, morbidity, and mortality in infants and young children. For many reasons, a vaccine that would prevent this disease is sought.

Plasmodium falciparum and Plasmodium vivax, the most common and severe forms of malaria, have host and stage specific proteins that can induce immunity to disease caused by this pathogen. Surprisingly, vaccines against stages that infect mosquitos will prevent the spread of malaria (transmission-blocking). We have developed a vaccine composed of a single protein, denoted as Pfs25, to induce transmission-blocking antibodies in the human host. These transmission-blocking antibodies will be ingested by the mosquito and inactivate the sexual forms of the plasmodia (ookinetes) as they develop in the midgut of the mosquito. Because Pfs25 is present only in the mosquito, humans do not develop antibody to this antigen even in endemic areas. No antibodies were detected against Pfs25, a 21-kD protein expressed on zygotes and ookinetes of P. falciparum and known to be a sensitive target of transmission-blocking antibodies. Theoretically, frequent boosting with this antigen, as is required for the other experimental malarial vaccines, would be necessary.

Our investigational vaccine is based upon the following:

1. Pfs25 is a low molecular weight protein and a poor immunogen.

   Bharti et al showed the protective action of antibodies to Pvs25 raised by intensive immunization of rabbits and mice (these regimes are not suitable for humans) to the recombinant protein. These findings have been confirmed;
2. Transmission of Plasmodia to mosquitos is mediated by their ingestion of gametocytes in the human bloodstream.

   Within 10 minutes, these gametocytes transform into gametes in the midgut of the mosquito. The male gametocyte fertilizes the female to form a zygote. Twenty four hours later ookinetes pierce the epithelium of the midgut and differentiates into an oocyst. This cell type forms the sporozoite that lodges in the salivary gland and is the infective form injected by the mosquito into the human host. Pfs25 may also be involved in survival of the ookinete in the midgut and its transformation into the oocyst;
3. The immunogenicity of poor immunogens is increased, especially in infants, by covalently binding them to medically-acceptable carrier proteins to form conjugates.

The Pfs25 was bound to itself by the synthetic scheme used for Haemophilus influenzae type b and other polysaccharides to proteins. The resultant conjugate was immunogenic and, unexpectedly, antibodies elicited by this vaccine continued to rise 3 months and 7 months after the second and third injections. The property of the Pfs25 conjugate to elicit long-lived antibody at high levels is unique to this construct. Our data from Pfs25 conjugate in mice suggest that administration of this vaccine to the whole population including infants along with their routine immunizations may be sufficient to elicit long-lived, effective transmission-blocking activity.

Our plan is to evaluate clinical lots of this conjugate for P. falciparum and for P. vivax, for their safety and immunogenicity in adults, children and infants, and then to establish a clinical site to test their efficacy.

ELIGIBILITY:
* ELIGIBILITY AND EXCULUSION CRITERIA

Healthy adults, 18 to 49 years of age of either sex who do not have any of the following conditions will be eligible to participate:

1. A chronic or progressive disease requiring chronic medication,
2. History of surgical splenectomy or abnormal immune system,
3. History of neurological symptoms or signs, or mental illness,
4. Anaphylactic shock following administration of any vaccine or any other severe allergic reaction.,
5. Women who are pregnant or intend to become pregnant during the vaccine study,
6. Had malaria or received a malaria vaccine previously,
7. Allergy to vaccine components or to nickel and yeast,
8. Had cancer, HIV/AIDS, Hepatitis B or C, Guillain Barre Syndrome, chronic skin disease or have abnormal liver functions or blood counts.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08-20; Primary Completion 2013-03-05 (Actual); Study Completion 2013-03-05 (Actual)

PRIMARY OUTCOMES:
Antibody

SECONDARY OUTCOMES:
Transmission-blocking activity

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Ying C Lin, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)

REFERENCES:
- [Background] Snow RW, Guerra CA, Noor AM, Myint HY, Hay SI. The global distribution of clinical episodes of Plasmodium falciparum malaria. Nature. 2005 Mar 10;434(7030):214-7. doi: 10.1038/nature03342. PMID 15759000
- [Background] Fernando SD, Gunawardena DM, Bandara MR, De Silva D, Carter R, Mendis KN, Wickremasinghe AR. The impact of repeated malaria attacks on the school performance of children. Am J Trop Med Hyg. 2003 Dec;69(6):582-8. PMID 14740872
- [Background] Carter R, Mendis KN, Miller LH, Molineaux L, Saul A. Malaria transmission-blocking vaccines--how can their development be supported? Nat Med. 2000 Mar;6(3):241-4. doi: 10.1038/73062. No abstract available. PMID 10700212